CLINICAL TRIAL: NCT01238588
Title: The Effect(s) of Sevelamer Carbonate (Renvela) on Atherosclerotic Plaque Inflammation Judged by FDG-PET Scan
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study stopped due to lack of funding.
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Kambiz Zandi-Nejad, MD, Instructor in Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010P002213
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Results first posted 2017-06-21 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Dialysis; Cardiovascular Disease; Atherosclerosis; Inflammation; Hyperphosphatemia
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Inflammation; Hyperphosphatemia | interventions — Sevelamer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sevelamer Carbonate (Renvela) (Other): Sevelamer Carbonate (Renvela). Information including those from the scans and blood test will be compared before and after treatment with Renvela.
  Interventions: Drug: Sevelamer Carbonate (Renvela)

INTERVENTIONS:
Drug: Sevelamer Carbonate (Renvela) — Patients' will be given doses of Renvela equivalent to their prior dose of calcium based phosphate binders and the dose will be titrated as necessary to achieve phosphate levels recommended by KDOQI guidelines.
  Other Names: Sevelamer carbonate; Renvela

SUMMARY:
The hypothesis is that switching calcium based phosphate binders to sevelamer carbonate will be associated with less inflammation including less atherosclerotic plaque inflammation (inflammation of the vessel walls).

ELIGIBILITY:
Inclusion Criteria:

* A signed consent form;
* Male or Female, 50 years or older;
* Diagnosed with end stage renal disease (ESRD), on maintenance hemodialysis for at least three (3) months;
* On calcium-based phosphate binders;
* Subject must be able to understand and provide informed consent;
* No known contraindications to therapy with sevelamer carbonate.

Exclusion Criteria:

* Any patient with a medical condition or taking any medications that would be contraindicated with the use of sevelamer carbonate, such as history of bowel obstruction;
* History of severe allergic reactions to the study medication;
* History of active infection (other than a simple respiratory tract infection) or acute gouty attack within 2 weeks prior to enrollment;
* Known serological positivity for Human Immunodeficiency Virus (HIV), Hepatitis B surface Antigen (HBsAg), or Hepatitis C Virus Antibody (HCV Ab) except dose with normal liver function tests (AST, ALT, Bilirubin, and Alkaline Phophatase) and no history of cirrhosis;
* Elevation of liver function tests at time of entry (Aspartate Aminotransferase (AST) and/or Alanine Aminotransferase (ALT) > 2 times the upper limit of normal);
* History of drug, alcohol, or chemical abuse within 6 months prior to enrollment;
* History of malignancy except those adequately treated, has completed treatment and clinically in remission for more than 6 month; adequately treated in-situ cervical carcinoma, or adequately treated basal or squamous cell carcinoma of the skin;
* History of an inflammatory disease such as systemic lupus erythematosus (SLE), rheumatoid arthritis or ulcerative colitis except those in remission for more than 6 months;
* Patients currently on sevelamer carbonate or sevelamer chloride or history of taking them for more than a week in the past three months;
* Patients receiving chronic anti-inflammatory therapy;
* Patients in whom FDG-PET/CT dual scans are contraindicated.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-06-10 (Actual); Primary Completion 2016-04-08 (Actual); Study Completion 2016-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kambiz Zandi-Nejad, MD, Principal Investigator — Brigham and Women's Hospital
Locations (10):
- United States (10):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Fresenius Boston-TKC, Boston, Massachusetts
  - BWH/FH/DCI Outpatient Dialysis Unit, Boston, Massachusetts
  - Fresenius Framingham (#1109), Framingham, Massachusetts
  - Fresenius Marlborough (#3448), Marlborough, Massachusetts
  - Fresenius Medford Dialysis (#1246), Medford, Massachusetts
  - Fresenius Quincy (#1610), Quincy, Massachusetts
  - Fresenius Roxbury (#1630), Roxbury, Massachusetts
  - DCI Dialysis Unit-Somerville, Somerville, Massachusetts
  - Fresenius QCDC-Weymouth (#9144), Weymouth, Massachusetts

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 24 patients enrolled in the study by signing the consent form of which 12 started the study. The other 12 never started the study due to various reasons (eg voluntary withdrawal, termination due to infection, transplant).
Period: Overall Study
Arm/Group | Sevelamer Carbonate (Renvela)
Started | 12
Completed | 9
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Sevelamer Carbonate (Renvela)
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Changes in Fluorodeoxyglucose (FDG)-Positron Emission Tomography (PET): FDG-PET/CT Dual Scan Score
Time Frame: Baseline and 6 months
Population: Scans were done but not analyzed due to early study termination (per funding source).
Arm/Group | Sevelamer Carbonate (Renvela)
Number analyzed (Participants) | 0
Value | 0

2. Primary Outcome: Changes in High Sensitivity C-Reactive Protein (Hs-CRP) Level
Time Frame: Baseline and 6 months
Population: Blood samples were collected but the measurements were not done due to early study termination (per funding source).
Arm/Group | Sevelamer Carbonate (Renvela)
Number analyzed (Participants) | 0
Value | 0

3. Primary Outcome: Changes in Interleukin-6 (IL-6) Level
Time Frame: Baseline and 6 months
Population: Blood samples were collected but the measurements were not done due to early study termination (per funding source).
Arm/Group | Sevelamer Carbonate (Renvela)
Number analyzed (Participants) | 0

4. Secondary Outcome: Albumin Levels
Time Frame: Baseline and 6 months
Population: Clinical lab data for this outcome measure was not collected from the medical record (for research purpose) due to early termination of the study (per funding source)
Arm/Group | Sevelamer Carbonate (Renvela)
Number analyzed (Participants) | 0
Value | 0

5. Secondary Outcome: Erythropoiesis Stimulating Agent (ESA) Dose Requirement
Time Frame: Baseline and 6 months
Population: Data for this outcome measure was not collected from the medical record due to early termination of the study (per funding source).
Arm/Group | Sevelamer Carbonate (Renvela)
Number analyzed (Participants) | 0
Value | 0

6. Secondary Outcome: Hemoglobin Level
Time Frame: Baseline and 6 months
Population: as for outcome 4
Arm/Group | Sevelamer Carbonate (Renvela)
Number analyzed (Participants) | 0
Value | 0

7. Secondary Outcome: Rate of Cardiovascular Events
Time Frame: Baseline and 6 months
Population: as for outcome 5
Arm/Group | Sevelamer Carbonate (Renvela)
Number analyzed (Participants) | 0
Value | 0

8. Secondary Outcome: Hemodialysis Access Stenosis/Thrombosis
Time Frame: Baseline and 6 months
Population: as for outcome 5
Arm/Group | Sevelamer Carbonate (Renvela)
Number analyzed (Participants) | 0
Value | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Sevelamer Carbonate (Renvela)
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sevelamer Carbonate (Renvela) (N=12)
Constipation (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrollment was much slower than anticipated due to logistical reasons, study at the direction of funding source terminated early and therefore none of the collected samples were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes